CLINICAL TRIAL: NCT00897143
Title: Isolation and Identification of Lung Cancer Precursor Cells From Malignant Pleural Effusion Specimens
Brief Title: Identifying Early Lung Cancer Cells in Malignant Pleural Effusion Samples From Patients With Primary Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI Left
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE1507; P30CA043703 (NIH); CASE1507 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: non-small cell lung cancer; malignant pleural effusion; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant; Small Cell Lung Carcinoma | interventions — Microarray Analysis; Flow Cytometry; Immunologic Techniques

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Malignant pleural effusion specimens from patients with primary lung cancer obtained from the Pathology Department at the University Hospitals of Cleveland.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: microarray analysis — analyzed using an immunomagnetic bead enrichment assay to isolate cells of epithelial origin
Genetic: mutation analysis — analyzed using an immunomagnetic bead enrichment assay to isolate cells of epithelial origin
Other: flow cytometry — analyzed using an immunomagnetic bead enrichment assay to isolate cells of epithelial origin
Other: immunologic technique — analyzed using an immunomagnetic bead enrichment assay to isolate cells of epithelial origin

SUMMARY:
RATIONALE: Studying samples of pleural fluid in the laboratory from patients with lung cancer may help doctors identify early lung cancer cells. It may also help the study of lung cancer in the future.

PURPOSE: This laboratory study is looking at malignant pleural effusion samples from patients with primary lung cancer to see if early lung cancer cells can be identified.

DETAILED DESCRIPTION:
OBJECTIVES:

* Isolate and identify lung cancer precursor cells in discarded pleural fluid specimens obtained during routine thoracentesis procedures for the diagnosis and treatment of malignant pleural effusions.

OUTLINE: Malignant pleural effusion specimens obtained from the Pathology Department at the University Hospitals of Cleveland are analyzed using an immunomagnetic bead enrichment assay to isolate cells of epithelial origin. The isolated cells are then stained with fluorescent DNA binding dye, Hoechst 33342, and other markers (i.e., CD133, CD24/CD44) and sorted by flow cytometry into progenitor and nonprogenitor subpopulations. The sorted subpopulations are separated and examined functionally by in vitro and in vivo studies. Sphere culture studies are also performed on the sorted subpopulations. The specimens may also be utilized for transcriptional profiling studies, RNAi studies, and for the establishment of long-term cultures and cell lines. DNA is also isolated and stored from tumor and nonepithelial normal cell compartments for future genetic studies on known and unidentified genetic abnormalities contributing to the development of lung cancer, such as EGFR, ErbB2, K-ras, and p53 mutational status.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically positive malignant pleural effusion secondary to primary small cell or non-small cell lung cancer
* Recruited from the Division of Hematology/Oncology, the Multidisciplinary Thoracic Oncology Group of Ireland Cancer Center, or the inpatient or outpatient units of Case Medical Center-University Hospitals

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Malignant pleural effusion samples from patients with primary lung cancer.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Isolation and identification of lung cancer precursor cells in malignant pleural effusion specimens

CONTACTS AND LOCATIONS:
Overall Officials: Balazs Halmos, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States